CLINICAL TRIAL: NCT00141583
Title: The Renin-Angiotensin System in Essential Hypertension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient accrual rate
Sponsor: St George's, University of London (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: LREC 01.87.10
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2007-05

CONDITIONS: Hypertension
Keywords: Renin-angiotensin system; ACE Inhibitor; Angiotensin Receptor Blocker
MeSH Terms: conditions — Hypertension | interventions — Enalapril; candesartan

INTERVENTIONS:
Drug: Enalapril 20 mg bd
Drug: Candesartan 8 mg bd

SUMMARY:
Although ACE Inhibitors and Angiotensin Receptor Blockers are effective blood pressure lowering agents, the exact mechanisms by which these agents lower BP are still not fully understood. This study aims to compare the blood pressure and hormonal responses (plasma renin activity and aldosterone) to the ACE inhibitor enalapril and ARB candesartan in individuals with mild essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Essential Hypertension
* SBP 140-159 mmHg
* DBP 90-99 mmHg

Exclusion Criteria:

* Intolerance of or allergy to ACE Inhibitors or ARBS
* Pregnant or Breastfeeding
* Pre-menopausal women
* Uncontrolled cardiac or renal failure
* Diabetes mellitus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2004-04; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change in BP
Change in PRA and aldosterone

CONTACTS AND LOCATIONS:
Overall Officials: Timothy WR Doulton, BSc MRCP, Principal Investigator — SGUL
Locations (1):
- Blood Pressure Unit, Dept. Cardiac & Vascular Sciences, SGUL, London, United Kingdom